CLINICAL TRIAL: NCT00137007
Title: A Multicenter, Open Label Trial Evaluating Intravenous Azithromycin Plus Intravenous Ampicillin/Sulbactam Followed by Oral Azithromycin Plus Intravenous Ampicillin/Sulbactam for the Treatment of Hospitalized Subjects With Community-Acquired Pneumonia (CAP)
Brief Title: Zithromax EV in Community-Acquired Pneumonia (CAP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0661082
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Azithromycin; sultamicillin

INTERVENTIONS:
Drug: Azithromycin
Drug: Ampicillin/sulbactam

SUMMARY:
The intravenous (IV) regimen containing azithromycin (Zithromax) plus ampicillin-sulbactam is consistent with current guidelines for the treatment of CAP. In fact the International guidelines for the treatment of CAP in hospitalised patients suggests the use of a combination between a b-lactam and a macrolide.

This trial will allow investigators to evaluate the efficacy of azithromycin plus ampicillin-sulbactam in the treatment of hospitalized subjects with community acquired pneumonia. In addition, this trial will allow investigators to evaluate the safety and toleration of combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must require hospitalization and intravenous therapy.
* Subjects must have a Fine pneumonia score > 70 (Fine Class > II).
* Subjects must have a medical history and clinical and radiological findings consistent with a community-acquired bronchopneumonia or lobar pneumonia. The following criteria must be met:

  * new infiltrate(s) on chest X-ray; AND
  * at least two of the CAP signs or symptoms.

Exclusion Criteria:

* Treatment with any systemic antibiotic for 24 hours or longer within 72 hours of the baseline visit, or treatment for more than 7 days within 15 days.
* Specific systemic diseases or other medical conditions that would interfere with the evaluation of the therapeutic response or safety of the study drug, including:

  * Known acquired immunodeficiency syndrome (AIDS) or suspected Pneumocystis carinii pneumonia;
  * Neutropenia;
  * Cavitary lung disease by chest X-ray;
  * Primary lung cancer or other malignancy metastatic to the lung;
  * Aspiration pneumonia;
  * Empyema;
  * Known or suspected tuberculosis;
  * Neoplastic disease;
  * Cystic fibrosis;
  * A history of any form of epilepsy or seizure;
  * DDM;
  * Bronchiectasis, bronchial obstruction or history of post-obstructive pneumonia (this does not exclude patients with chronic obstructive pulmonary disease);
  * Significant gastrointestinal or other conditions which may affect study drug absorption; and
  * Significant cardiovascular disorders.
* Immunosuppressive therapy, defined as chronic treatment with known immunosuppressant medications
* Impaired hepatic function, as shown by, but not limited to, AST, (SGOT), or ALT (SGPT) greater than three times the laboratory upper limit of normal, or total bilirubin greater than two times the upper limit of normal.
* Subjects already hospitalized or who resided in a long-term-care facility for greater than 14 days before the onset of symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2003-11; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical efficacy of intravenous (IV) azithromycin 500 mg once daily plus IV ampicillin/sulbactam 3 grams twice a day (BID) for 2 to 5 days
followed by oral azithromycin 500 mg once daily plus IV ampicillin/sulbactam 3 grams.

SECONDARY OUTCOMES:
To evaluate the eradication of baseline pathogens of IV azithromycin plus IV ampicillin/sulbactam followed by oral azithromycin plus IV ampicillin/sulbactam at Visit 3 and Visit 4

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer